CLINICAL TRIAL: NCT06608654
Title: The New Application of Electronic Endoscope in the Visual Diagnosis and Treatment of Intrauterine Fetal Distress During Labor
Brief Title: Application of Electronic Endoscope in Fetal Distress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Taixing People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EEFD-01
Record Dates: First submitted 2024-08-12; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Fetal Distress; Fetal Hypoxia
MeSH Terms: conditions — Fetal Distress; Fetal Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fetal distress (Experimental)
  Interventions: Device: endoscope application

INTERVENTIONS:
Device: endoscope application — Intrauterine bronchoscopy application for fetal distress during labor

SUMMARY:
Fetal distress is a common emergency in obstetrics, which refers to the combined symptoms of fetal health and life in utero due to acute or chronic hypoxia, with an incidence of 2.7% to 38.5%. Fetal distress is mainly related to abnormal amniotic fluid, umbilical cord entanglement and compression, which is an important reason for the increase of cesarean section rate during delivery. At present, the diagnosis of fetal distress mainly relies on electronic monitoring of fetal heart, and the false positive rate is high. Intrauterine pressure catheter has not been widely used because of the little effect of intrauterine treatment and the increase of infection. Endoscopy has been widely used in the diagnosis and treatment of various specialties at present, but the diagnosis and treatment during childbirth are still in a blind area. The characteristics of endoscopic visualization provide a new idea for the diagnosis and treatment of fetal distress during delivery, especially for the etiological diagnosis and treatment of umbilical cord factors. The use of intraauterine endoscope during delivery can make up for the defects of intrauterine pressure catheter, realize the visual diagnosis of the causes of fetal distress such as oligoamniotic fluid, meconium contamination of amniotic fluid, umbilical cord compression caused by entangling and true junction, etc. At the same time, it can also improve the intrauterine environment by perfusion of saline for the causes of fetal embarrassment, correct fetal distress, and extend the observation time during labor. It is beneficial to reduce caesarean section during labor.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 20-45 years with single pregnancy;
2. Intrauterine fetal distress occurs during labor (during the first stage of labor), and the fetal membrane was already broken;
3. Fetal heart monitoring category II, after stopping oxytocin, oxygen inhalation, change of position, intravenous fluid and other measures can not improve;
4. Understand the research procedures, be able to follow the procedures of the research protocol, and voluntarily sign a written consent.

Exclusion Criteria:

1. Type III fetal heart monitoring for pregnant women who require emergency c-section
2. Pregnant women with GBS positive
3. Pregnant women suspected of chorioamniotic infection
4. Pregnant women have signs of reproductive system infection (vaginal inflammation, cervicitis, uterine infection)
5. Pregnant women suspected of uterine rupture
6. Pregnant women with abnormal contractions: excessive strong contractions
7. Check the fetus for serious deformities during pregnancy
8. Check pregnant women with serious abnormal functions of cardiovascular system, urinary system, digestive system, reproductive system and other organs

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
fetal distress rate | through study completion, an average of 1 year
  fetal distress rate during first stage of labor

SECONDARY OUTCOMES:
vaginal delivery rate | through study completion, an average of 1 year
  baby was deliverd vaginally
Incidence of maternal infection | through study completion, an average of 1 year
  materna infection was diagnozed up to 42 days after delivery
Neonatal asphyxia rate | through study completion, an average of 1 year
  Neonatal asphyxia was diagnozed after the baby was deliverd
neonatal NICU admission rate | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No